CLINICAL TRIAL: NCT05596708
Title: A Single-arm, Forward-looking, Exploratory Clinical Study of Telitacicept in Patients With Refractory IgA Nephropathy
Brief Title: Study of Telitacicept in Patients With Refractory IgA Nephropathy
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SZNK
Record Dates: First submitted 2022-10-25; First posted 2022-10-27 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2022-10

CONDITIONS: IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — telitacicept

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telitacicept treated group (Experimental)
  Interventions: Drug: Telitacicept

INTERVENTIONS:
Drug: Telitacicept — Telitacicept will be subcutaneously injected at a dose of 240mg per week, lasting for 104 weeks.

SUMMARY:
The goal of this clinical trial is to explore the effectiveness and safety of Telitacicept in adults with refractory IgA nephropathy.

The main questions it aims to answer are:

* To evaluate the clinical efficacy of Telitacicept in patients with refractory IgA nephropathy.
* To evaluate the safety and adverse reaction of Telitacicept in patients with refractory IgA nephropathy.

Participants will be subcutaneously injected with 240mg of Telitacicept once per week.

Study subject: After 6 months of sequential treatment with renin-angiotensin system (RAS) blockers or glucocorticoids, patients with pathological biopsy of 0.7≥5 g/24 hours of proteinuria was confirmed as refractory IgA nephropathy.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form.
2. IgA nephropathy was confirmed by pathological biopsy.
3. Age range: ≥ 18 years old, ≤ 70 years old, male or female.
4. During the screening period, the 24-hour urine protein of Visit 1 and Visit 2 should meet at least one ≥0.75g/24h, and the 24-hour urine protein ≥ 0.75g/24h at Visit 3.
5. Measured glomerular filtration rate or estimated GFR (using the CKD-EPI formula) > 35 mL/min/1.73 m2.
6. Participants had received a basic regimen including ACE inhibitors/ARBs for 12 weeks prior to randomization, and the dose of ACE inhibitors/ARBs (within the maximum tolerated range) was stable for 4 weeks prior to randomization.

Exclusion Criteria:

1. Abnormal laboratory indicators of participants need to be excluded.
2. Secondary IgA nephropathy need to be excluded.
3. Specific pathologic or clinical renal disease types, and IgA nephropathy that may require hormone therapy.
4. Patients who have experienced any of the following cardiovascular and cerebrovascular events within the 12 weeks prior to screening.
5. Use of systemic corticosteroids within 3 months prior to randomization (except local, nasal inhalation, etc.)
6. Immunosuppressants were used within 3 months prior to randomization.
7. Patients requiring hospitalization for active infection or intravenous anti-infective therapy within 3 months prior to randomization.
8. Previously or currently diagnosed active tuberculosis Untreated latent tuberculosis.
9. Herpes zoster HIV antibody positive or HCV antibody positive during the screening period.
10. Those who currently have active hepatitis or have severe liver disease and medical history.
11. Patients with malignant tumors.
12. Pregnant and lactating women, and men or women with planned children during the trial period.
13. Those who could not avoid the use of nephrotoxic drugs during the trial.
14. Allergic to human biological products.
15. Patients who have been given any of the clinical trial drugs 4 weeks prior to randomization or within 5 times the half-life of the experimental drug (whichever is longer).
16. Patients deemed ineligible for the trial by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Complete clinical response | 3-year
  a. Proteinuria: protein-to-creatinine ratio <0.2; b. Stable renal function: eGFR decreased by less than 5ml/min/1.73m2 from baseline at the end of the 3-year trial phase.
The absolute value of eGFR | 3-year
  The absolute value of eGFR decreased by more than 15 ml/min/1.73m2 over 3 years from baseline
Changes in 24-hour urinary protein | 104 weeks
  Changes in 24-hour urinary protein at week 104 compared with baseline.

SECONDARY OUTCOMES:
eGFR decrease | 3-year
  The estimated glomerular filtration rate (eGFR) decreased by more than 30 ml/min/1.73 m2 from baseline.
Need for dialysis | 3-year
  progression to end-stage renal disease

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided